CLINICAL TRIAL: NCT02793401
Title: A Comparison of the Efficacy of High Intensity Laser and Ultrasound Therapies in Patients With Chronic Shoulder Pain: A Randomized Controlled Single Blind Study
Brief Title: Chronic Shoulder Pain Treatment: High Intensity Laser or Ultrasound
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Burcu Metin Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BursaYIERH
Record Dates: First submitted 2016-05-20; First posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Shoulder Pain Chronic
Keywords: High Intensity Laser; Ultrasound; Chronic Shoulder Pain
MeSH Terms: interventions — Ultrasonography; Transcutaneous Electric Nerve Stimulation; Exercise Therapy; Balneology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HILT group (Active Comparator): 71 of the patients were in the HILT group
  Interventions: Device: Hıgh İntensity Laser (HILT); Device: Hotpack; Device: Transcutaneous electrical nerve stimulation; Other: Therapeutic exercises; Other: Balneotherapy
- US Group (Active Comparator): 70 of the patients were in the US group.
  Interventions: Device: Ultrasound; Device: Hotpack; Device: Transcutaneous electrical nerve stimulation; Other: Therapeutic exercises; Other: Balneotherapy

INTERVENTIONS:
Device: Hıgh İntensity Laser (HILT) — HILT was performed using a BTL-6000 High Intensity Laser, 12 W(watt), 1064 nm device was a hot laser with Nd: YAG LASER source. In HILT group, the investigators applied the device on the shoulder area in two phases: phase I - analgesia, and phase II - biostimulation.
  Arms: HILT group
Device: Ultrasound — BTL 4710 US device was applied at 3 MHz frequency, and 1.5watt/cm2 intensity over 25 cm2 surface area. Headpiece area of the device was 5 cm2, and the application was performed as the head of device was positioned at 90º (perpendicular) at full contact for 5 minutes by using gel, and performing continuous circular motions.
  Arms: US Group
Device: Hotpack — All patients had the same physical therapy (PT) protocol including hot pack (HP) for 20 min/session,
Device: Transcutaneous electrical nerve stimulation — All patients had the same physical therapy (PT) protocol includingTENS (Fizyotens 4000, Fizyomed Medical Devices Ltd,Turkey) (50-100 Hz) for 20 min/session,
  Other Names: TENS
Other: Therapeutic exercises — All patients had the same physical therapy (PT) protocol including therapeutic exercises for shoulder muscles
Other: Balneotherapy — All patients had the same physical therapy (PT) protocol including balneotherapy in 38-40 °C thermomineralized water for 20 minutes.

SUMMARY:
The investigators aimed to evaluate the short-term efficacy of High Intensity LASER Therapy (HILT) and Ultrasound (US) treatment in chronic shoulder pain. It's a prospective, randomized, controlled, single blind study.141 patients were randomized into two groups, as HILT (n=71) and US (n=70) groups. HILT or US treatment was applied to the patients in addition to 14 sessions of Hotpack (Hp) + Balneotherapy + Exercise treatment. Pre-treatment (Pre-T), Post-treatment 1st day (Post-T1st day) and Post-T findings for the 30th day (Post-T 30th day) were recorded using the visual analog scale (VAS) and shoulder pain and disability index (SPADI) scoring.

DETAILED DESCRIPTION:
Chronic shoulder pain, which negatively affects the quality of life due to pain and loss of functions, is the third most common painful condition of the musculoskeletal system[1] The aim of the study was to determine more effective conventional physical treatment method (HILT or US) for pain and daily activities of patients with chronic shoulder pain which was difficult to treat, and had unfavorable effects on patient life quality. This prospective, randomized, controlled, single blind study was conducted at the Physical Treatment and Rehabilitation Training and Research Hospital and ethics board approval was obtained.A total of 210 patients, who presented to the hospital with chronic shoulder pain, were evaluated for inclusion in the study. Patients to be included in the study were divided into two groups by the investigating physician, using simple randomization, and their treatment was organized. Forms detailing the patients' (demographics, VAS scores and SPADI) were completed by another investigating physician who was blind to the type of treatment the patients would receive. The same investigating physician completed Post-treatment 1st day (Post-T1st day) and Post-T findings for the 30th day (Post-T 30th day) forms and recorded the data. Patients who were randomly divided into two groups received treatment for two weeks (14 days) are shown below:

* Group 1: Hotpack (HP)+ Balneotherapy+ Exercise + HILT
* Group 2: Hotpack (HP)+ Balneotherapy+ Exercise + US

Patients in both groups received HP to the affected shoulder region for 20 minutes and balneotherapy, in mineral water pool at 38-400C for 20 minutes, for seven consecutive days. ROM exercises and Codman exercises, in a level not to increase the severity of the pain of the patient, were given and stretching and strengthening exercises were taught to the patients.The patients performed these exercises daily in two sets with five repeats in each set.

HILT was performed using a BTL-6000 High Intensity Laser, 12 W(watt), 1064 nm device was a hot laser with Nd: YAG LASER source. BTL 4710 US device was applied at 3 MHz frequency, and 1.5watt/cm2 intensity over 25 cm2 surface area. Headpiece area of the device was 5 cm2, and the application was performed as the head of device was positioned at 90º (perpendicular) at full contact for 5 minutes by using gel, and performing continuous circular motions. Patients were evaluated using VAS and SPADI in pre-treatment (Pre-T), Post-T1st day and Post-T 30th day.

ELIGIBILITY:
Inclusion Criteria:

* The presence of shoulder pain for more than 3 months patients.

Exclusion Criteria:

* Limitation in the shoulder movements of more than 20%,
* Receiving physical therapy and injection treatment to the same shoulder region in the previous year,
* Malignancy,
* The presence of radicular pain and cervical myofascial pain syndrome,
* A history of acute trauma,
* A prior history of fracture in the shoulder to be treated,
* A prior history of surgical intervention and implantation of a metal implant to the affected shoulder,
* Inflammatory rheumatoid disease.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
VAS | Change from Baseline in VAS scores at 15 days and 45 days
  Patients were evaluated using by visual analog scale(VAS) in pre-treatment (Pre-T), 15th day and 45th day. VAS is a frequently used test worldwide, for which reliability and safety studies have been performed.
SPADI | Change from Baseline in SPADI scores at 15 days and 45 days.
  Patients were evaluated using SPADI in pre-treatment (Pre-T), 15th day and 45th day. SPADI was developed to measure shoulder discomfort. Its evaluation includes two parts: pain and disability. Part 1 includes five questions in the pain subgroup and measures the pain experienced by the patient over the previous week using VAS (0 no pain, to 10,most severe pain). Part 2 is the disability subgroup and includes eight questions and measures the degree of difficulty (0 no difficulty, to 10, requires help) in the movements of the patient during the last week. SPADI includes 13 questions, and zero point refers to maximal well-being and 130 points refers to maximal sickness.The investigators evaluated each part of the SPADI (shoulder pain index (SPI), shoulder disability index (SDI) and total SPADI) separately.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Metin Ökmen, MD, Study Director — Bursa Yuksek Ihtisas Education and Research Hospital; Korgün Ökmen, MD, Principal Investigator — Bursa Yuksek Ihtisas Education and Research Hospital; Kağan Özkuk, MD, Study Chair — Abant İzzet Baysal Physical Therapy and Rehabilitation Education and Research Hospital; Bilal Uysal, MD, Study Chair — Abant İzzet Baysal Physical Therapy and Rehabilitation Education and Research Hospital; Refia Sezer, MD, Study Chair — Abant İzzet Baysal Physical Therapy and Rehabilitation Education and Research Hospital; Engin Koyuncu, MD, Study Chair — Ankara Physical Therapy and Rehabilitation Education and Research Hospital
Locations (1):
- Bursa Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Bursa, Turkey (Türkiye)